CLINICAL TRIAL: NCT00273117
Title: Transnasal and Conventional Oral Diagnostic Gastroscopy. A Prospective Randomised Study.
Brief Title: Transnasal and Oral Gastroscopy.
Status: Terminated | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Other Study IDs: MC-01-GLO; Ethics commitee nr KA00066m
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2006-01

CONDITIONS: Upper Gastrointestinal Disease, Duodenal or Gastric Ulcer.
Keywords: transnasal gastroscopy; tachycardia; hypoxemia
MeSH Terms: conditions — Gastrointestinal Diseases; Stomach Ulcer; Tachycardia; Hypoxia

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

INTERVENTIONS:
Procedure: transnasal gastroscopy

SUMMARY:
Two groups of patients were randomised into two groups of either transnasal gastroscopy or conventional type gastroscopy (n=98). The aim of the study was to evaluate the cardiorespiratory effects and sideeffects of the two methods, and to evaluate the technical features of the transnasal endoscope.

DETAILED DESCRIPTION:
Introduction Esophagogastroduodenoscopy is the gold standard investigation for upper gastrointestinal disorders. To make the procedure safer and more comfortable, thinner endoscopes for conventional oral or for transnasal intubation have been designed. Several trials have been conducted suggesting greater patient tolerance with the thinner scope. At the same time scope features have improved and are increasingly compatible with the standard endoscope. This prospective, randomised study was conducted to evaluate the cardiopulmonary effects, the patient tolerance, and endoscopist evaluation comparing thin transnasal with conventional transoral endoscopy.

Patients and Methods Outpatients referred to diagnostic, upper gastrointestinal endoscopy were included consecutively after written informed consent. Inclusion criteria were age over 18 years, Danish-language, no history of disease in the nasal cavity and intended diagnostic endoscopy. Ninety-eight patients were included and randomised to either conventional oral gastroscopy (OG) or transnasal gastroscopy (TG).The patients were randomized by consecutively numbered envelopes.

The patients answered a questionnaire clarifying their previous experience of gastroscopy, and if relevant, the discomfort of previous examination and their anxiety for the actual examination on a visual analogue scale (VAS scale). A post endoscopy questionnaire evaluated discomfort during the examination in general, during introduction of the endoscope and for the rest of the examination (VAS scale). The following parameters were assessed by answering yes or no; gagging, choking, pain from the nose, throat and the stomach. The patients stated whether the degree of discomfort had been greater, lesser or as expected compared to previous endoscopy and whether they in a future gastroscopy would prefer sedation, and finally they stated their preference for a future procedure (OG/TG).

TG were carried out using Olympus Videoscope GIF-N230 (Olympus Optical Ltd., Tokyo, Japan) with an outer diameter of 6 mm and working length of 925 mm (first 15 patients); and later Olympus Videoscope GIF-XP160 (33 patients) with an outer diameter of 5.9 mm, and a working length of 1030 mm. OG were carried out using Olympus Videoscope GIF-Q160 with an outer diameter of 9.5 mm and a working length of 1030 mm.

All patients received topical anaesthesia; before TG xylocain gel were inhaled into each nostril and before OG xylocain spray (10 mg/dose), 4 doses were spayed into the pharyngeal cavity. Intravenous sedation using midazolam were used only if specifically requested by the patient. The patients were positioned in the left lateral recumbent position during the procedures. Endoscopies were performed by experienced endoscopists.

Arterial oxygen saturation (SpO2 ) and heart rate (HR) were measured by a pulse oximeter (Nellcor Symphony N-3000, Nellcor Puritan Bennet Inc., Pleasanton, CA) twice with an interval of one minute before the procedure; twice during the procedure (one and three minutes after intubation) and finally one and two minutes after extubation. The minimum SpO2 and maximum HR were noted as was the duration of the procedure. Biopsies were taken when indicated, and the qualities of the biopsies were assessed. Adverse effects during the endoscopies were noted; e.g. epistaxis.

After the endoscopy, the endoscopists answered a questionnaire evaluating the following parameters using a VAS score: intubation, ability to aspirate gastric contents, visualization of the esophagus, the stomach, the bulb and the second part of duodenum. The presence of chromatic aberrations (after flushing and aspiration), were also assessed. It was noted whether the length of the scope was sufficient, and also in case of TG, the presence of uni- or bi-lateral stenosis of the nasal cavity and looping in esophagus. If TG could not be carried out, the reasons were noted.

Finally, the endoscopists assessed their total subjective evaluation of the endoscopy on a one-to-six scale (one: unacceptable, six: perfect).

ELIGIBILITY:
Inclusion Criteria:

* diagnostic gastroscopy, written informed consent

Exclusion Criteria:

* history of broken nose or disease of the nasal cavity, no Danish language, age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-02; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Merete Christensen, MD, Principal Investigator — Dept. of Cardiothoracic Surgery, Copenhagen University Hospital Rigshospitalet, Denmark
Locations (1):
- Dept of Surgery University Hospital of Glostrup, Glostrup Municipality, Glostrup, Denmark